CLINICAL TRIAL: NCT04251715
Title: A Phase II Study of Induction Systemic mFOLFIRINOX Followed by Hepatic Arterial Infusion of Floxuridine and Dexamethasone Given Concurrently With Systemic mFOLFIRI as a First-Line Therapy in Patients With Unresectable Liver-Dominant Intrahepatic Cholangiocarcinoma
Brief Title: mFOLFIRINOX Followed by Hepatic Arterial Infusion of Floxuridine and Dexamethasone With Systemic mFOLFIRI for Unresectable Liver-dominant Intrahepatic Cholangiocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Skye C Mayo, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016033; NCI-2020-00477 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016033 (Other: OHSU Knight Cancer Institute); HELIX-1 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Liver and Intrahepatic Bile Duct Carcinoma; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIA Intrahepatic Cholangiocarcinoma AJCC v8; Stage IIIB Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Floxuridine; 5-fluoro-2'-deoxyuridine; Irinotecan; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- mFOLFIRINOX, Floxuridine-DEX, mFOLFIRI (Experimental): Treatment Period 1 - mFOLFIRINOX for 4 cycles (cycle = 14 days) Cycle 1
  * Oxaliplatin 85 mg/m2 intravenously (iv) over 2 hours
  * Folinic acid 400 mg/m2 iv over 2 hours
  * Irinotecan 165 mg/m2 iv over 90 minutes
  * Fluorouracil 400 mg/m2 iv bolus after folinic acid
  * Fluorouracil 2,400 mg/m2 continuous infusion over 46 hours
  Dosages on Cycle 2, 3, and 4 will be reduced by 25% Treatment Period 2 - HAI delivery of floxuridine + mFOLFIRI for 2 cycles (cycle = 28 days)
  * Floxuridine-DEX (with heparin and saline) - 0.12 mg/kg/day; via HAI pump, adjusted for weight and flow rate
  mFOLFIRI on Day 15
  * Irinotecan 180 mg/m2 iv over 30 minutes to 1 hour
  * Folinic acid 400mg/m2 iv over 30 minutes to 1 hour
  * 5-FU 1000 mg/m2 continuous infusion over 46 hours
  Interventions: Drug: Dexamethasone; Drug: Floxuridine; Device: Implanted Medical Device; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Dexamethasone — Given intraarterially via HAI pump
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Floxuridine — Given intraarterially via HAI pump
  Other Names: 2''-Deoxy-5-fluorouridine; 5-Fluoro-2''-deoxyuridine; 5-Fluorodeoxyuridine; 5-Fluorouracil deoxyriboside; 5-FUdR; FDUR; Floxuridin; Fluorodeoxyuridine; Fluorouridine Deoxyribose; Fluoruridine Deoxyribose; FUdR; WR-138720
Device: Implanted Medical Device — Implanted hepatic arterial infusion pump by surgical oncology, to deliver HAI therapy
  Other Names: IMPLANTED
Drug: Irinotecan — Given IV
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the efficacy and safety of systemic induction of mFOLFIRINOX, followed by hepatic arterial infusion (HAI) floxuridine-dexamethasone administered concurrently with systemic mFOLFIRI in treating patients with liver-dominant intrahepatic cholangiocarcinoma (ICC) that cannot be removed by surgery (unresectable). Drugs used in chemotherapy regimens, such as mFOLFIRINOX and mFOLFIRI (Oxaliplatin, Irinotecan, Fluorouracil, Folinic acid, Floxuridine) work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Delivering chemotherapy via HAI (hepatic arterial infusion) can allow for liver-directed treatment while limiting toxic side effects typically seen with traditional chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the toxicity, safety and tolerability of hepatic arterial infusion (HAI) floxuridine therapy.

II. Evaluate the efficacy of systemic induction of oxaliplatin, leucovorin calcium (folinic acid), irinotecan hydrochloride, and fluorouracil (modified [m] FOLFIRINOX), followed by HAI of floxuridine-dexamethasone (DEX) administered concurrently with systemic irinotecan hydrochloride, leucovorin calcium (folinic acid), and fluorouracil (mFOLFIRI).

SECONDARY OBJECTIVES:

I. To evaluate tumor response to treatment and participant survival. II. Assess rate of post-operative complications. III. Evaluate serious post-operative complications following surgical placement of the HAI pump.

EXPLORATORY OBJECTIVES:

I. To assess the radiographic response using diffusion weighted imaging (DWI) as part of an magnetic resonance imaging (MRI) examination.

II. Determine whether, compared to historical controls, induction mFOLFIRINOX combined with integrated HAI of floxuridine-DEX and systemic mFOLFIRI treatment will improve patient quality of life (QoL) including fatigue and depression.

III. Investigate molecular signature associated with intrahepatic cholangiocarcinoma (ICC).

IV. Generate a differential expression pattern of ribonucleic acid (RNA)s (microRNA [miR] and messenger RNA [mRNA]) in patients with ICC derived from tumor samples compared to adjacent normal liver samples as well as lymphatic tissue, blood and bile).

V. Characterize the changes in the population of circulating hybrid cells (CHCs) pre-, during, and post-treatment.

OUTLINE: This is a phase II, single arm, study that consists of a two-part treatment plan (Treatment Periods 1 and 2) of systemic induction of mFOLFIRINOX, followed by HAI floxuridine-DEX administered concurrently with systemic mFOLFIRI. The first 6 patients enrolled will be part of a safety run-in, after which enrollment could be expanded to additional 24.

After laparoscopic staging, eligible patients will receive a systemic regimen of mFOLFIRINOX with 25% dose reduction of oxaliplatin, irinotecan, and fluorouracil administered every 2-weeks for 4 cycles (8 weeks) (Treatment Period 1). After completing mFOLFIRINOX induction, participants' disease will be re-evaluated by MRI/CT imaging. Only those that achieve disease control based on RECIST criteria (v1.1) will be eligible for HAI therapy via a laparotomy and placement of a HAI pump. (Treatment Period 2).

After completing 2 cycles of HAI treatment with concurrent FOLFIRI, participants will undergo repeat MRI/CT imaging to assess disease response. An image-guided liver biopsy will be performed after completion of the 8 weeks of treatment of HAI floxuridine/dexamethasone combined with systemic mFOLFIRI of Treatment Period 2. Optional extrahepatic biopsies may be collected from participants demonstrating disease progression. Participants with controlled disease (as defined by RECIST criteria) may receive additional cycles of HAI-delivered floxuridine and dexamethasone, along with systemic administration of mFOLFIRI. Completion of QoL questionnaires and interviews will take place at baseline, at the end of treatment period 1 and prior to each HAI treatment cycle, and again at the end of study, and again from the End of Study up to 24 months post study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed intrahepatic cholangiocarcinoma (ICC; also variously reported as peripheral cholangiocarcinoma, cholangiolar carcinoma or cholangiocellular carcinoma) with confirmation of the pathologic diagnosis at Oregon Health & Science University (OHSU)
* Surgically unresectable liver-dominant ICC, or multifocal ICC considered surgically unresectable or resection is contraindicated

  * For liver-dominant ICC, disease must comprise < 70% of the liver parenchyma, as defined by computed tomography (CT) liver segmental volumetrics
* Limited extrahepatic disease

  * Clinical or radiographic evidence of metastatic disease to regional lymph nodes and limited extrahepatic disease to the lungs is permitted at the discretion of the principal investigator (PI)
* Radiographically measurable hepatic disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria
* Disease must be considered technically unresectable at the time of preoperative evaluation or radiographically multifocal as determined by hepatobiliary surgical oncologists
* Participants should be treatment naive. Those previously treated with systemic chemotherapy (e.g., gemcitabine, cisplatin, or other investigational agents) may be eligible at the discretion of the PI
* Participants with an Eastern Cooperative Oncology Group (ECOG) 0 or 1 status (Karnofsky >= 60), and can be considered candidates for general anesthesia, abdominal exploration and hepatic artery pump placement
* Participants with treated chronic hepatitis (e.g., treated hepatitis B virus [HBV], treated hepatitis C virus [HCV]) are eligible, but must be Child-Pugh class A
* White blood cell (WBC) >= 3000 cells/mm^3
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3
* Platelet count >= 100,000/mm^3
* International normalized ratio (INR) =< 1.5
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR creatinine clearance >= 40 ml/min (> 0.675 ml/sec) using Cockcroft-Gault equation
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Participants must be able to read, understand, and sign informed consent
* Participants must be willing and able to fully comply with required post-operative visits associated with HAI chemotherapy

Exclusion Criteria:

* Presence of extensive or multifocal metastatic extrahepatic or peritoneal disease. Clinical or radiographic evidence of metastatic disease to regional lymph nodes will be allowed, as will limited pulmonary disease at the discretion of the OHSU PI
* Prior treatment with floxuridine, oxaliplatin, or irinotecan
* Prior treatment with hepatic arterial infusion therapy
* Known to have experienced an allergic reaction or other signs of intolerance to implanted devices
* Body size that is insufficient to accommodate the physical size of the pump
* Diagnosis of sclerosing cholangitis
* Diagnosis of hepatic encephalopathy
* Clinical evidence of portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis) or hepatic venous wedge pressures > 8 mmHg if available
* History of multiple abdominal operations that would preclude HAI pump placement
* Active infection
* Current biliary obstruction requiring placement of endoscopic or transhepatic stents for biliary decompression
* Presence of aberrant or replaced hepatic arterial anatomy not amenable to placement of a hepatic arterial infusion pump catheter as judged by the operating surgeon
* History of peripheral neuropathy > grade 1
* Allergies to iodine contrast medium, that cannot be premedicated with steroids per institutional radiology guidelines (e.g., dexamethasone)
* Uncontrolled severe coagulation disorders (INR > 1.5 in patients not on warfarin therapy)
* Pregnant or lactating women
* History of malignancy other than cholangiocarcinoma within 5 years prior to screening, with the exception of:

  * Malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival [OS] rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, melanoma in situ, localized prostate cancer, ductal carcinoma in situ, or
  * Stage I uterine cancer or a malignancy whose natural history or treatment has, in the opinion of the principal investigator, the potential to interfere with the safety or efficacy assessment of the intervention under investigation
* Life expectancy =< 12 weeks
* Inability to comply with study and/or follow-up procedures
* Emotional or psychiatric problems that would preclude successful participation in the hepatic arterial infusion program as judged by the one of the study investigators, and further corroborated by the mandatory interview and assessment with medical oncology social worker
* EXCLUSION CRITERIA FOR TREATMENT PERIOD 2
* Participants with radiographic evidence of extrahepatic disease
* Evidence of extrahepatic disease found at laparoscopy during open surgical exploration for HAI pump implantation. Participants with extrahepatic disease found at time of laparoscopy or laparotomy will not undergo surgical placement of HAI pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of abnormal liver function | Up to 2 years
  Defined by unacceptable elevation in liver enzymes, or radiographic evidence of biliary sclerosis on computed tomography (CT)/magnetic resonance imaging (MRI) (as measured following the completion of 2 cycles of hepatic arterial infusion [HAI] in Treatment Period 2).
Disease control rate (DCR) - during HAI+SYS | Up to 2 years
  DCR is defined as the percentage of patients who have achieved complete response (CR), partial response (PR), or stable disease (SD). Measured from beginning of Treatment Period 2 to end of Treatment Period 2 during treatment with HAI + systemic chemotherapy (SYS).

SECONDARY OUTCOMES:
DCR - entire treatment | Up to 2 years
  Measured from beginning of Treatment Period 1 to end of Treatment Period 2 (i.e., from the beginning of the entire treatment protocol until the end).
DCR - FOLFIRINOX | Up to 1 year
  Measured from beginning of Treatment Period 1 to end of Treatment Period 1 (i.e., during the treatment with oxaliplatin, irinotecan, and fluorouracil [FOLFIRINOX] alone).
Progression free survival (PFS) - FOLFIRINOX | Up to 1 year
  Measured from beginning of Treatment Period 1 to end of Treatment Period 1 (i.e., during the treatment with FOLFIRINOX alone).
PFS | Up to 2 years
  Measured from beginning of Treatment Period 2 to up to 1 year after the end of Treatment Period 2 (i.e., during the treatment with HAI floxuridine + irinotecan hydrochloride and leucovorin calcium [folinic acid] [modified(m)FOLFIRI].
Overall response rate (ORR) | Up to 2 years
  Measured from beginning of Treatment Period 1 to end of Treatment Period 2 (i.e., from the beginning of the entire treatment protocol until the end).
Overall survival (OS) | Up to 2 years
  Measured at the end of Treatment Period 1, at the end of Treatment Period 2, and at 1 year, and the whole study period.
Proportion of liver toxicity in participants receiving HAI floxuridine + dexamethasone therapy | Up to 1 year
Incidence of serious post-operative complications | Up to 9 weeks after surgery
  Defined as complications occurring within 9 weeks following surgery and >= grade III per the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Skye C Mayo, MD, MPH, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542